CLINICAL TRIAL: NCT02622815
Title: Hypercoagulation Screening as Innovative Tool for Risk Assessment, Early Diagnosis and Prognosis in Cancer
Brief Title: Hypercoagulation Screening in Cancer
Acronym: HYPERCAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other); Istituto Neurologico Mediterraneo Neuromed S. R. L (Other); Fondazione Humanitas per la Ricerca (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); ASL Roma 1 (Unknown); Istituti Ospedalieri Bergamaschi Srl (Other); ASST Bergamo Ovest (Other); Istituti Tumori Giovanni Paolo II (Network)
Responsible Party: Principal Investigator, ANNA FALANGA, Director of the Division of Immunohematology and Transfusion Medicine, Papa Giovanni XXIII Hospital
Other Study IDs: AIRC5xmille - 12237
Record Dates: First submitted 2015-11-24; First posted 2015-12-07 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy Blood Donors; Moli-sani Subjects; Cancer Patients
Keywords: Hypercoagulation; Thrombosis; Cancer Risk Assessment; Cancer Prognosis
MeSH Terms: conditions — Thrombophilia; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma, serum and tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy blood donors: 10,000 highly controlled blood donors in the age range 30-70 years
- Moli-sani subjects: A sample of 1,000 tumor cases have been identified so far and samples from these participants will be analyzed compared to 1,000 controls from randomly extracted from the Moli-sani cohort (parent cohort).
- Cancer patients: 4,000 Patients with breast, lung, and gastrointestinal tumors.

SUMMARY:
There is a complex, mutual relationship between cancer and thrombosis. Indeed, the tumor has the capacity to activate the hemostatic system and this leads to an increased thrombotic risk in cancer patients. Even in the absence of clinical manifestations, cancer patients are commonly characterized by hemostatic abnormalities, recognized only by laboratory testing, which define the 'hypercoagulable state'. Of interest, hypercoagulation has been repeatedly reported to be associated with tumor progression and poor prognosis in various carcinomas. On the other hand, thrombotic event can represent the first signal of the presence of an occult tumor. These findings suggest that the coagulant pathway might play a role in the preclinical phase of cancer. The investigators hypothesize that a persistent, subclinical activation of the hemostatic system in an otherwise healthy subject, may predispose not only to thrombosis, but also to tumor formation and spreading. A major problem in primary cancer prevention is the lack of effective predictive markers of the disease. The HYPERCAN is an ongoing prospective Italian multicenter study organized around two tightly-interconnected research programs aiming to: 1_the assessment of thrombotic markers as a tool for cancer risk prediction in two large populations of healthy subjects, i.e. a group of healthy blood donors of Bergamo and Milano Provinces and a subgroup of Moli-sani subjects of the Molise region; and 2_ the evaluation whether thrombotic markers and/or the occurrence of overt thrombosis (or disseminated intravascular coagulation) may be prognostic of cancer disease outcomes (i.e. overall survival, progression free survival in metastatic cancer, disease free survival in limited disease) in cancer patients with different types of solid tumors (i.e. breast, lung and gastrointestinal cancers).

Therefore, the assessment of cancer risk occurrence in healthy individuals might be useful for anticipation of cancer diagnosis. In addition, the results of this study might help to evaluate whether thrombotic markers may be prognostic of cancer outcomes independently of the disease extension.

ELIGIBILITY:
Blood donors_

Inclusion Criteria:

* good health
* signed informed consent.

Exclusion Criteria: (considering 10-15 days from blood sampling)

* inflammations/infections/fever;
* recent vaccinations;
* recent surgery;
* anticoagulant therapy.

Cancer patients_

Inclusion Criteria:

* with life expectation higher than 3 months;
* patients with breast, lung or gastrointestinal tumors candidated for chemotherapy regimen;
* ECOG PS 0-2;
* adeguate bone marrow and renal function;
* signed informed consent.

Exclusion Criteria:

* acute medical illness;
* terminal conditions or life expectancy less than 3 months;
* under low molecular weight heparin at therapeutic dosage.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Blood donors (age range 30-70 years), who agree to participate, fulfill a specific questionnaire on their lifestyle and donate venous blood samples at the enrollment into the study, and after 6-12 months.
  The parental cohort of the Moli-sani project included 24,325 subjects (>35 years) from the Molise region. Blood samples have been collected and stored in the Moli-sani biobank available to this project.
  Cancer patients of both genders (>18 years) with new diagnosis of non small cell lung cancer, gastrointestinal tumors, and breast cancer are enrolled at different recruiting sites. Blood samples are collected at the enrollment and at specific time points during follow-up without interfering with clinical management.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2012-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of blood donors with a diagnosis of cancer | within 5 years from the date of the enrollment
  Samples collected from identified participants with cancer diagnosis will be assessed to determine the hypercoagulation profile (ratio for laboratory analysis cancer case : healthy control from same cohort = 1:3, matched for age and gender)
Incidence of Thrombotic events among enrolled cancer patients | within 5 years from the date of the enrollment
  Identification of cancer patients with evidence of thrombotic event derived from review of clinical records.

SECONDARY OUTCOMES:
Incidence of Cancer progression among enrolled cancer patients | within 5 years from the date of the enrollment
  Identification of cancer patients with evidence of cancer progression derived from review of clinical records.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Falanga, MD, Principal Investigator — A.O. Papa Giovanni XXIII - Recruiting
Locations (8):
- Italy (8):
  - Istituti Ospedalieri Bergamaschi S.r.l. - Policlinico San Marco, Osio Sotto, Bergamo
  - A.S.S.T. Bergamo Ovest, Treviglio, Bergamo
  - I.R.C.C.S. Istituto Neurologico Mediterraneo NEUROMED, Pozzilli, Isernia
  - Fondazione Humanitas per la Ricerca, Rozzano, Milan
  - Papa Giovanni XXIII Hospital - Oncology Unit, Bergamo
  - Papa Giovanni XXIII Hospital - S.I.M.T., Bergamo
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - ASL Roma 1 - ACO San Filippo Neri & San Giovanni Maria Addolorata Hospital, Rome